CLINICAL TRIAL: NCT06946225
Title: A First-in-human, Open-label Trial to Evaluate the Combination of ACTengine® IMA203 With mRNA-4203 in Previously Treated, Unresectable or Metastatic Cutaneous Melanoma or Synovial Sarcoma Patients (ACTengine® IMA203-102)
Brief Title: ACTengine® IMA203 Combined With mRNA-4203
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Immatics US, Inc. (Industry)
Collaborators: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMA203-102
Record Dates: First submitted 2025-04-19; First posted 2025-04-27 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Cutaneous Melanoma; Synovial Sarcoma
Keywords: immunotherapy; T-cell therapy; cutaneous melanoma; synovial sarcoma; RNA vaccine; Immatics; Moderna
MeSH Terms: conditions — Melanoma; Sarcoma, Synovial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IMA203 with mRNA-4203 in participants with metastatic cutaneous melanoma or synovial sarcoma (Experimental): This is a non-comparative, open-label trial with different cohorts investigating IMA203 in combination with mRNA-4203.
  Interventions: Biological: IMA203; Biological: mRNA-4203

INTERVENTIONS:
Biological: IMA203 — Following non-myeloablative chemotherapy for lymphodepletion (LD) with fludarabine (FLU) and cyclophosphamide (CY), participants will receive a single infusion of IMA203 on Day 1 and adjunctive therapy with low dose interleukin (IL)-2 for up to 10 days, starting approximately 24 h after IMA203 infusion.
  Other Names: anzutresgene autoleucel; anzu-cel
Biological: mRNA-4203 — mRNA-4203 will be administered starting on Day 15 after IMA203 infusion at the earliest. mRNA-4203 will be given for 12 cycles (28 day cycle length); during Cycle 1 it will be given on Day 1 and Day 15 and in Cycles 2-12 it will be given on Day 1.
  Other Names: anzu-cel

SUMMARY:
This purpose of this clinical trial is to evaluate the safety, tolerability and anti-tumor activity of IMA203 in combination with different doses of mRNA-4203. The trial includes participants with previously treated unresectable or metastatic cutaneous melanoma (CM) or synovial sarcoma (SS).

DETAILED DESCRIPTION:
This clinical trial is a multi-center, open-label, non-comparative Phase 1 a/b trial to assess the safety, tolerability, and anti-tumor activity of the combination of IMA203 and mRNA-4203 in HLA-A*02:01 positive patients with previously treated, unresectable or metastatic cutaneous melanoma (CM) and synovial sarcoma (SS).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed and documented cutaneous melanoma (CM) or synovial sarcoma (SS) with unresectable or metastatic disease
* HLA-A*02:01 positive
* Adequate selected organ function per protocol
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
* Life expectancy more than 5 months
* CM participants who must have disease progression (resistance, toxicity) on or after at least one PD-1 inhibitor
* SS participants must have received (or declined) at least one line of treatment (including SoC) and are still in need of further systemic therapy.
* Female participants of childbearing potential must use adequate contraception prior to trial entry until 12 months after the infusion of IMA203 and 15 days after the last mRNA 4203 dose administration

Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* History of other malignancies (except for adequately treated basal or squamous cell carcinoma or carcinoma in situ) within the last 3 years
* Pregnant or breastfeeding
* Serious autoimmune disease
* History of cardiac conditions as per protocol
* Prior allogenic stem cell transplantation or solid organ transplantation
* Concurrent severe and/or uncontrolled medical disease that could compromise participation in the study
* History of hypersensitivity to cyclophosphamide, fludarabine, or IL-2
* History of hypersensitivity to mRNA-based medicines
* Positive for HIV infection or with active hepatitis B virus (HBV) or active hepatitis C virus (HCV) infection
* Any condition contraindicating leukapheresis
* Participants with lactate dehydrogenase (LDH) greater than threshold allowed per protocol
* Participants with active brain metastases prior to lymphodepletion
* Concurrent treatment in another clinical trial or a device trial that could interfere with the IMA203 treatment
* Participants with renal impairment AND reduced bone marrow reserve per protocol

Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicities (DLTs) | one year post infusion of IMA203
  Number of DLTs will be used to determine the maximum tolerated dose (MTD) and/or recommended dose for extension (RDE) after treatment with IMA203 product in combination with mRNA-4203
Number of treatment emergent adverse events (AEs), AEs of special interest, serious AEs (SAEs), changes in laboratory parameters and vital signs, and frequency of dose interruptions, reductions and discontinuations | one year post infusion of IMA203
  Used to evaluate safety and tolerability of treatment with IMA203 in combination with mRNA-4203

SECONDARY OUTCOMES:
Objective response rate (ORR) | one year post infusion of IMA203
  complete response (CR) and partial response (PR) based on best overall response (BOR), locally assessed using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Duration of response (DOR) | one year post infusion of IMA203
  CR and PR, locally assessed using RECIST v1.1
Disease control rate (DCR) | one year post infusion of IMA203
  CR, PR and stable disease (SD) lasting 6 or more weeks following the infusion of IMA203, locally assessed using RECIST v1.1
Progression-free survival (PFS) | one year post infusion of IMA203
  locally assessed using RECIST v1.1
Concentration of IMA203 transgene in peripheral blood | one year post infusion of IMA203
  Evaluate the pharmacokinetics of T-cell receptor (TCR) engineered T cells in combination with mRNA-4203

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of California San Francisco, San Francisco, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas